CLINICAL TRIAL: NCT05886335
Title: Evaluation of the Influence of Timing of Post-transplant Cyclophosphamide in Allogeneic Haematopoietic Stem Cell Transplant Patients.
Brief Title: Influence of Timing PTCy in AlloSCT
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-CFM-2023-45
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Cyclophosphamide Toxicity; Allogenic Haematopoetic Transplantation
Keywords: haemorrhagic cystitis; cyclophosphamide; allogenic haematopoetic transplantation
MeSH Terms: conditions — Cystitis, Hemorrhagic | interventions — Cyclophosphamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cystitis hemorrhagic: Cystitis hemorrhagic grade II-III
  Interventions: Drug: Cyclophosphamide
- Non Cystitis hemorrhagic: Non cystitis hemorrhagic or grade I
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — Time of administration

SUMMARY:
Cyclophosphamide, administered after the infusion of haematopoietic progenitor cells, is used to prevent graft-versus-recipient disease (GVHD) in patients undergoing allogeneic haematopoietic stem cell transplantation (allogeneic HSCT) and has been shown to reduce the incidence of GVHD.

Cyclophosphamide can cause haemorrhagic cystitis as a result of the direct toxicity of its metabolite acrolein to the bladder mucosa or urothelium upon accumulation in the urine. Hyperhydration and the administration of mesna, which forms a non-urotoxic compound with acrolein, are among the most commonly used strategies to prevent this. The administration of cyclophosphamide in the morning is also recommended.

The protocol for post-transplant cyclophosphamide states that it should be started at least 72 hours (days +3 and +4) after haematopoietic progenitor infusion, but this interval can be extended to 84 hours (day +3.5). After reviewing the recommendations to reduce the risk of haemorrhagic cystitis, it was recommended to delay the infusion of cyclophosphamide to the early morning of days +4 and +5, although in reality, taking into account the hours since the infusion of haematopoietic progenitors, it would be days +3.5 and +4.5 instead of days +3 and +4 in the afternoon/evening. This change will mean a delay of 12 hours in the start of cyclophosphamide, so the investigators will refer to day +3.5 from the infusion of the haematopoietic precursors.

DETAILED DESCRIPTION:
Cyclophosphamide administered after haematopoietic stem cell infusion is used for the prevention of graft-versus-recipient disease (GVHD) in patients undergoing allogeneic haematopoietic stem cell transplantation (allo-SCT) and has been shown to reduce the incidence of GVHD.

However, cyclophosphamide can cause haemorrhagic cystitis (HC) as one of the best known adverse effects. This is due to the direct toxicity of the cyclophosphamide metabolite, acrolein, to the bladder mucosa or urothelium as it accumulates in the urine. The incidence of HC can vary from 10 to 70% of patients and increases the number of days spent in hospital as well as morbidity and mortality after transplantation. Among the most common risk factors and causative agents, in addition to cyclophosphamide, are BK polyomavirus infections, with cyclophosphamide-induced HC often occurring within 72 hours of the administration of cyclophosphamide.

There are several strategies to prevent cyclophosphamide-induced HC, such as hyperhydration with saline and forcing diuresis with furosemide, alkalinisation of diuresis or administration of mesna, which forms a non-urotoxic complex with acrolein in the urinary tract and prevents tissue damage. However, further studies are needed to understand the best strategy to prevent HC, especially in the setting of allo-SCT.

In order to ensure proper hydration, to promote diuresis during the day and to reduce the time that acrolein is in contact with the mucosa, the administration of cyclophosphamide in the morning is recommended.

There are several strategies to prevent cyclophosphamide-induced HC, such as hyperhydration with saline and forcing diuresis with furosemide, alkalinisation of diuresis or administration of mesna, which forms a non-urotoxic complex with acrolein in the urinary tract and prevents tissue damage. However, further studies are needed to understand the best strategy to prevent HC, especially in the setting of allo-SCT.

In order to ensure proper hydration, to promote diuresis during the day and to reduce the time that acrolein is in contact with the mucosa, the administration of cyclophosphamide in the morning is recommended.

The usual protocol for the administration of cyclophosphamide (PTCy) after transplantation states that it should be started at least 72 hours (days +3 and +4) after the infusion of haematopoietic progenitors, but this interval can be extended to 84 hours (days +3.5) and the days of administration have been changed to days +3 and +5 with optimal results. In some patients, the infusion of haematopoietic precursors is carried out in the afternoon because of the need for nursing care. This meant that cyclophosphamide had to be administered in the evening, 72 hours after the infusion of the precursors. After review of the recommendations to reduce the risk of haemorrhagic cystitis, it was recommended that cyclophosphamide infusion be delayed in the morning on days +4 and +5, although in reality, taking into account the hours since haematopoietic progenitor infusion, these would be days +3.5 and +4.5 instead of days +3 and +4 in the afternoon/evening. This change means a 12-hour delay in the start of cyclophosphamide. Therefore, the investigators refer to day +3.5 from the infusion of haematopoietic progenitors.

ELIGIBILITY:
Inclusion Criteria:

* Adult recipients (>18 years old) of Allo-SCT
* Allo SCT between January 1, 2014 and December 31, 2022
* PTCy dose 50 mg/kg x 2 days

Exclusion Criteria:

* Patients with no record of time of administration of PTCy
* PTCy dose of 30 mg/kg x 2 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received cyclophosphamide after haematopoietic progenitor transplantation, consecutively, at the HSCSP, between January 2014 and December 2022.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
incidence haemorrhagic cystitis Grade II-IV | 6 months
  To compare the incidence of grade II to IV haemorrhagic cystitis, according to the CTCAE classification, depending on the schedule of post-transplant cyclophosphamide administration in consecutive patients.

SECONDARY OUTCOMES:
GVHD acute and chronic | 6 months
  To compare the incidence of acute and chronic graft-versus-host disease.
Mortality and relapsed | 6 months
  To compare the incidence of transplant-related mortality and recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided